CLINICAL TRIAL: NCT04069000
Title: Implementing a Mindfulness-informed, Evidence-based Social and Emotional Program With Kindergarten Students Within a Trauma-informed Framework
Brief Title: Mind Up (MindUP) Evaluation With Grade 3 Students
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We collected pre-intervention data but the COVID-19 pandemic and resulting school closures ended the intervention; thus post-intervention data were not collected. Our funding window has closed and we will not recommence this study.
Sponsor: Western University, Canada (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Claire Crooks, Professor; Director, Centre for School Mental Health, Western University, Canada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0000039458
Record Dates: First submitted 2019-08-12; First posted 2019-08-28 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Child Development
Keywords: Social-Emotional Learning; Classroom Climate; Self-concept; Academic Skills

STUDY DESIGN:
Intervention Model Description: Children within grade 3 classrooms will be evaluated in one of three conditions. One condition includes classrooms that will implement MindUP with students for the first time. A second condition includes classrooms that will implement MindUP, but has students who have largely been exposed to MindUP every year since kindergarten. The third condition is the comparison group wherein classroom teachers will deliver their usual curriculum and teaching strategies.
Masking Description: Due to the nature of the intervention (i.e., classroom teachers both implement the program (or not) and provide ratings of students' behaviour, it is not feasible to have blinded conditions. Most school-based prevention programs of this type are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular grade 3 classrooms (Active Comparator): Students in this condition will participate in the regular grade 3 program. Educators will use their usual teaching methods to meet educational outcomes, including standards for social-emotional learning.
  Interventions: Behavioral: Regular grade 3 program
- First time MindUP participants (Experimental): Students in this condition will participate in MindUP for the first time. Their classroom teachers will receive training and implement the program during the school year.
  Interventions: Behavioral: Mindfulness-based social-emotional learning program
- Repeat MindUP participants (Experimental): Students in this condition are in schools where MindUP has been implemented since they were in kindergarten (although some students may not have participated in those first three years, depending on when they moved to the school). Their classroom teachers will receive training and implement the program during the school year.
  Interventions: Behavioral: Mindfulness-based social-emotional learning program

INTERVENTIONS:
Behavioral: Mindfulness-based social-emotional learning program — Grade 3 teachers implement MindUP in their classrooms over the academic year. MindUP is a manualized program informed by cognitive-developmental neuroscience, contemplative science, positive psychology, and social-emotional learning. The curriculum consists of 15 sequential lessons taught in 10-15 minute chunks and cross-curricular extension activities. There are four lesson units: Getting Focused (introduction to brain structure and function, the core practice, and how focused awareness affects brains and feelings), Sharpening Your Senses (focus on internal experiences such as mindful smelling and tasting), It's All About Attitude (focus on cognitive experiences such as positive mindset, perspective-taking, and practicing gratitude), and Taking Action Mindfully (performing acts of kindness to others and building positive relationships). An essential component is the core practice, a focused breathing exercise and mindfulness practice that is implemented three times daily.
  Other Names: MindUP
  Arms: First time MindUP participants; Repeat MindUP participants
Behavioral: Regular grade 3 program — Grade 3 teachers are expected to implement activities to achieve a number of pre-specified social-emotional learning outcomes that are identified by the Ministry of Education. Educators have leeway over how they achieve these curriculum expectations and they will report on a weekly basis regarding their implementation of social-emotional learning activities.
  Arms: Regular grade 3 classrooms

SUMMARY:
Mind Up (MindUP) is a mindfulness-based social-emotional learning program for children that has shown promising evidence of effectiveness across several domains (including executive functioning and behavioral symptoms). MindUP has exploded in popularity in recent years, but much of the existing research is limited by sample size, lack of accounting for clustering, or has been conducted by the program developers. In this study we are evaluating MindUP with grade three students (~age 8) in three conditions; students who receive MindUP for the first time (n=~150 in 8-10 classrooms), students have been receiving MindUP since kindergarten (~150 in 8-10 classrooms), and students in comparison classrooms (i.e., no intervention; ~150 students in 8-10 classrooms). Regular classrooms teachers will receive training in trauma-informed approaches and the MindUP program prior to implementing. Students will be assessed in the fall and at the end of the school year using structured rating scales; they will also provide self-report data. In November 2020, students' grade 4 teachers will provide another set of ratings to be used as 6-month follow-up data. The primary outcome is social-emotional learning. Secondary outcomes include executive functioning, academic skills, classroom climate, and self-concept.

DETAILED DESCRIPTION:
Study Design and Overview:

Social-emotional learning programs have a strong evidence base documenting their effectiveness. More recently, there has been increasing interest in social-emotional learning programs that include mindfulness; however, there is much less research on these programs, and much of the existing work has been hampered by small sample sizes. In this project, the investigators will examine the association between participation in the MindUP program and social-emotional outcomes in grade three students. The investigators are using a quasi-experimental design with pre-post data collection from students and educators. Students are nested in classrooms, and the clustered nature of the data will be accounted for in analyses. The study will identify changes in social-emotional behaviour, executive functioning, classroom climate, academic skills, and self-concept through a combination of teacher and self-report data using standardized scales.

Participants:

The investigators plan to recruit approximately 24 educators and 450 grade three students in approximately 24 classrooms. More or fewer classrooms will be recruited as needed to reach the intended sample size of 150 students in each of the three conditions.

Procedures:

The school district partnering on this project will identify 24 classrooms to participate. The first condition (~150 children in 8-10 classrooms) will participate in MindUP during the school year. The second condition (~150 children in 8-10 classrooms) includes children who have been participating in MindUP since kindergarten receiving the program in grade 3. The third group is a comparison condition where teachers will not implement the program. All implementing teachers will receive a half-day training on trauma-informed practice and a full-day training in MindUP before beginning the intervention.

Classroom teachers will send home consent forms for guardians to complete. Children will provide their own assent when the researchers come to classrooms to collect data. Surveys will be completed in October 2019 and again in May 2020. In November 2020, the students' grade 4 teachers will provide ratings for a 6-month follow-up.

To understand program implementation, educators will be asked to complete a brief online survey at the end of each week to report on their weekly engagement with MindUP lesson plans generally, and breathing breaks specifically. They will also be asked to report additional SEL activities. Educators in comparison classrooms will complete a weekly summary of their SEL learning activities as well.

Planned Analyses The primary comparisons will be between the group receiving MindUP for the first time versus the comparison groups (both immediately after intervention, and at 6-month follow-up). A secondary set of analyses will compare the group who have received MindUP for three years previously to the comparison group to see if they continue to make gains relative to the comparison group. Finally, we will also conduct moderator analyses using parent-reported adversity to test our hypothesis that students who have experienced more adversity will show greater gains.

ELIGIBILITY:
Inclusion Criteria:

* Decision to implement the MindUP program is made at the school level, with agreement from classroom teachers
* All students in a classroom in any of the three arms of the study are eligible to participate

Exclusion Criteria:

* Students with very low literacy or cognitive functioning may not be able to complete the self-report measures, but can still participate in the teacher-rating component of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Social and emotional learning | Change from baseline to post-intervention; one school year (approximately 6 months)
  Composite Social-Emotional Learning (SEL) score from the Social Skills Improvement System-Social Emotional Learning Edition (SSIS-SEL); the score is transformed from a raw score based on norms provided in the manual; higher scores are better. Scores are standardized with a mean of 100 and a standard deviation (SD) of 15.
Social and emotional learning (follow-up) | Change from baseline to 6-month follow-up; one calendar year
  Composite Social-Emotional Learning (SEL) score from the Social Skills Improvement System-Social Emotional Learning Edition (SSIS-SEL); the score is transformed from a raw score based on norms provided in the manual; higher scores are better. Scores are standardized with a mean of 100 and a standard deviation of 15.

SECONDARY OUTCOMES:
Academic skills | Change from baseline to post-intervention; one school year (approximately 6 months)
  Academic skills reported by teachers on SSIS-SEL and/or report card and standardized testing data. Higher scores are better.
Social and Emotional Learning Subscales | Change from baseline to post-intervention; one school year (approximately 6 months)
  Subscales from the SSIS-SEL (self-awareness; self management; social awareness; responsible decision-making; relationships); higher scores are better. Scores are standardized and norm-referenced with a mean of 100 and a standard deviation of 15.
Self-concept | Change from baseline to post-intervention; one school year (approximately 6 months)
  Child's view of themselves as assessed by the Feelings, Attitudes, and Behaviors Scale for Children (FAB-C). Higher scores are indicative of poorer functioning (i.e., feeling negative about oneself or feeling socially unaccepted). T scores are used to interpret the level of concerns as reported by children on the FAB-C. These scores are linear transformations of the raw scale scores (M = 50, SD = 10). T scores provide information about an individual's scores relative to the scores of respondents in the standardization sample. Percentiles represent the percentage of children in the standardization sample with scores at or below the same value. For all FAB-C subscales, T scores over 60 are considered somewhat elevated and T scores over 65 are considered significantly elevated.
Class climate | Change from baseline to post-intervention; one school year (approximately 6 months)
  Classroom cohesion and satisfaction as measured by the My Class Inventory-Short Form. Both cohesion and satisfaction are measured with six yes/no items, such that children can score between 0 and 6 on each subscale. If the two scales are moderately correlated (as expected give the age of the children), then we will sum them for one class climate scale (ranging from 0-12; higher scores indicate higher cohesion and satisfaction in the classroom).
Executive functioning | Change from baseline to post-intervention; one school year (approximately 6 months)
  General executive control deficits as measured by the Behavior Rating Inventory of Executive Function, Second edition (BRIEF-2). Higher scores are indicative of poorer functioning. T scores are used to interpret the level of executive functioning as reported by teachers on the BRIEF-2 rating forms. These scores are linear transformations of the raw scale scores (M = 50, SD = 10). T scores provide information about an individual's scores relative to the scores of respondents in the standardization sample. Percentiles represent the percentage of children in the standardization sample with scores at or below the same value. For all BRIEF-2 clinical scales and indexes, T scores from 60 to 64 are considered mildly elevated, and T scores from 65 to 69 are considered potentially clinically elevated. T scores at or above 70 are considered clinically elevated.
Executive functioning (follow-up) | Change from baseline to 6-month follow-up; one calendar year
  General executive control deficits as measured by the Behavior Rating Inventory of Executive Function, Second edition (BRIEF-2). Higher scores are indicative of poorer functioning. T scores are used to interpret the level of executive functioning as reported by teachers on the BRIEF-2 rating forms. These scores are linear transformations of the raw scale scores (M = 50, SD = 10). T scores provide information about an individual's scores relative to the scores of respondents in the standardization sample. Percentiles represent the percentage of children in the standardization sample with scores at or below the same value. For all BRIEF-2 clinical scales and indexes, T scores from 60 to 64 are considered mildly elevated, and T scores from 65 to 69 are considered potentially clinically elevated. T scores at or above 70 are considered clinically elevated.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Crooks, PhD, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — https://www.csmh.uwo.ca/research/mindup.html
- See also: MindUP program website — http://mindup.org